CLINICAL TRIAL: NCT00267111
Title: Local Anaesthesia [Topical Amethocaine Gel (Ametop)] for Intramuscular Injection in Term Neonates: A Randomized Controlled Trial.
Brief Title: Topical Amethocaine Gel for Intramuscular Injection in Term Neonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Striving for Excellence Fund, Mount Sinai Hospital (Unknown)
Responsible Party: Principal Investigator, Vibhuti Shah, Staff Neonatologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-0086-E; 00267111 (Registry Identifier: www.clinicaltrials.gov)
Record Dates: First submitted 2005-12-15; First posted 2005-12-20 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: Infant,newborn; Topical anesthesia; Intramuscular injection
MeSH Terms: conditions — Pain | interventions — eucerin; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amethocaine gel 4% Group (Experimental): 1 g of topical amethocaine gel 4%
  Interventions: Drug: Amethocaine gel 4%
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Eucerin plus

INTERVENTIONS:
Drug: Eucerin plus — 1g, single application
  Arms: Placebo Group
Drug: Amethocaine gel 4% — 1 g, single application
  Other Names: Ametop
  Arms: Amethocaine gel 4% Group

SUMMARY:
This study will examine the efficacy of topical amethocaine gel (Ametop) in decreasing the pain response in term neonates subjected to intramuscular injection for administration of vitamin K.

Study Hypothesis: We believe that topical amethocaine gel will be superior to placebo in decreasing the pain from intramuscular injection in term neonates.

DETAILED DESCRIPTION:
This randomized controlled trial will assess the efficacy of topical amethocaine gel (Ametop) compared with placebo (Eucerin plus) in decreasing the pain response in term neonates subjected to intramuscular injection for administration of vitamin K. Neonatal pain response between groups will be assessed using the Neonatal Facial Action Coding System (NFCS) which is currently the gold standard for infant pain assessment, latency to first cry and cry duration. Parents' (father) perception of infant's pain will be assessed using a visual analogue scale (VAS) when possible.

Neonates will be randomized to receive either amethocaine gel or identical appearing placebo administered locally at the injection site (the upper part of the neonate's thigh) using a pre-prepared syringe 30 minutes prior to the administration of vitamin K. The gel or placebo will be covered using a Saran wrap. Each neonate will be videotaped during the procedure. Parents (father) will be present during the procedure (observing) so that they (he) can assess their neonate's pain response using VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Term neonates > 37 weeks and
2. Birth weight > 2500 grams (appropriate for gestational age - AGA) -

Exclusion Criteria:

1. Neonates with major congenital anomalies
2. Neonates with known neurological abnormalities (antenatally diagnosed)
3. Neonates who require admission to the neonatal intensive care unit at birth

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2003-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vibhuti S Shah, MD, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Shah VS, Taddio A, Hancock R, Shah P, Ohlsson A. Topical amethocaine gel 4% for intramuscular injection in term neonates: a double-blind, placebo-controlled, randomized trial. Clin Ther. 2008 Jan;30(1):166-74. doi: 10.1016/j.clinthera.2008.01.018. PMID 18343253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between July 2003 and December 2004 in the Labour and Delivery Unit of Mount Sinai Hospital.
Groups:
- Placebo Group: 1 g Eucerin plus was used as a placebo.
Period: Overall Study
Arm/Group | Amethocaine Gel 4% Group | Placebo Group
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amethocaine Gel 4% Group | Placebo Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 55 | 110
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (1.1) | 39.2 (1.0) | 39.25 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 30 | 23 | 53
Region of Enrollment [Number; unit: participants]
  Canada | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Assessed by Neonatal Facial Action
Description: The presence or absence of 3 facial actions (brow bulge, eyes squeeze and deepening of the nasolabial furrow) were scored in 2 second intervals for the first 20 seconds (or less if the phase lasted < 20 seconds) of each procedure phase from the videotapes by a trained research assistant. The data were then collapsed for each facial action into the percentage of time the infant expressed the action. An overall pain score was computed by summing the percentage scores for the three facial actions and then dividing by three. The score ranged from 0% to 100% with higher values suggesting more pain.
Time Frame: For the purpose of analysis IM injection procedure was divided into 4 phases: baseline , cleansing, injection and recovery phases.. For each phase facial actions were scored for the first 20 seconds or less if the phase lasted < 20 seconds.
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: Percentage of time
Groups:
- 1 g Amethocaine Gel 4%: 1 g Amethocaine gel 4% was used as the active drug
Arm/Group | 1 g Amethocaine Gel 4% | Placebo Group
Number analyzed (Participants) | 54 | 53
Percentage of time
  Baseline | 14 (26) | 18 (28)
  Cleaning | 30 (39) | 44 (42)
  Injection | 70 (32) | 75 (34)
  Recovery | 79 (24) | 76 (28)
Statistical Analysis 1: Comparison: 1 g Amethocaine Gel 4% vs Placebo Group; We hypothesized that topical amethocaine gel 4% would reduce the pain from IM injection. The sample size was based on the pain scores obtained from a previous study that compared pain response during IM injection. To achieve a clinically significant reduction in pain scores by 20% between groups with 80% power and an alpha value of < 0.05, we estimated sample size of 49 neonates in each group. A total of 110 neonates were enrolled to account for possible dropouts and missing data; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Statistical analyses were performed using SPSS v12, USA). Pain scores were compared between groups by means of the Student t-test. A p-value of < 0.05 was considered significant

2. Secondary Outcome: Visual Analogue Scale
Description: Parents and nurses were asked to assess the infant's pain response during the procedure using Visual analogue scale (VAS) on an unmarked horizontal 10 cm continuous line where 0="no pain" on the left side and 10="worst possible pain" on the right side. Parents and nurses were trained to use the VAS prior to the IM injection.
Time Frame: During the entire procedure
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: Cms
Groups:
- Amethocaine Gel 4% Group: 1 g Amethocaine gel 4% was used as the active drug
Arm/Group | Amethocaine Gel 4% Group | Placebo Group
Number analyzed (Participants) | 54 | 55
Cms
  Parents VAS rating | 4.6 (2.3) | 4.6 (2.4)
  Nurses VAS rating | 5.0 (2.1) | 4.9 (2.3)
Statistical Analysis 1: Comparison: Amethocaine Gel 4% Group vs Placebo Group; We hypothesized that parents and nurses will report lower pain scores as assessed by visual analogue scale in topical amethocaine gel 4% compared to placebo group. This was a secondary outcome and no power calculation was performed; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Amethocaine Gel 4% Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 7/54 | 4/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amethocaine Gel 4% Group (N=54) | Placebo Group (N=53)
Local erythema (Skin and subcutaneous tissue disorders) | 7 (54) | 4 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No